CLINICAL TRIAL: NCT02759718
Title: Clinical Effectiveness of Serum Chromogranin A (CgA) Levels on Diagnostic Relevance, Response After Surgical Resection and Recurrence of Pancreatic Endocrine Tumors (PET)
Brief Title: Clinical Effectiveness of Serum Chromogranin A Levels on Diagnostic of Pancreatic Neuroendocrine Tumors
Acronym: CgA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Song Cheol Kim, professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CgA_PNET_AMC_Korea
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Non Functioning Pancreatic Endocrine Tumor
Keywords: pancreatic neuroendocrine tumor; chromogranin A
MeSH Terms: conditions — Non functioning pancreatic endocrine tumor; Adenoma, Islet Cell | interventions — Chromogranin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pancreatic neuroendocrine tumor (Experimental): chromogranin A
  Interventions: Biological: Chromogranin A

INTERVENTIONS:
Biological: Chromogranin A — The plasma level of chromogranin A (CgA) was measured in enrolled patients who was diagnosed as PNET in preoperative condition.After surgical resection, the CgA level was only measured in the the patient with PNET. In the PNET group, the CgA level was regularly checked in a 3, 6, 12, and 24 months after surgical resection.
  Other Names: CgA

SUMMARY:
Chromogranin A (CgA) is a glycoprotein with a molecular weight of 49 to 52 kDa produced by chromaffin cells of the adrenal medulla, enterochromaffin-like (ECL) cells, and endocrine cells of the stomach and pancreas, and it is the precursor to several functional peptides including vasostatin and pancreastatin.

Importantly, CgA can be measured in the serum or plasma or detected within the secretory vesicles as a general diagnostic biomarker for neuroendocrine tumors (NETs), and plasma CgA levels also provide information regarding tumor burden and response to treatment. It has a sensitivity and specificity between 27% and 81%.

Some studies have noted an association between CgA concentrations and tumor location or degree of differentiation. It has also been proposed that plasma CgA levels are more frequently elevated in well-differentiated tumors compared with poorly differentiated tumors of the midgut. Some other clinical series have provided evidence of an association between plasma CgA levels and the extent of disease, tumor burden, or presence of metastases, and high baseline levels of CgA are suggestive of a poor prognosis.

However, there exist still controversies the effectiveness of serum CgA levels on diagnostic relevance, treatment response after surgical resection or sandostatin analog, clinicopathologic features of pancreatic neuroendocrine tumors (PNETs).

To date, moreover, a precise association between CgA levels and survival has not been clearly demonstrated, although a number of studies suggest that this relationship may exist. There, especially, is no relevant data on value of serum CgA level for clinical usefulness in Korean population.

DETAILED DESCRIPTION:
An interventional, prospective, multi center pilot study to assess the clinical relevance of CgA levels in patients with PNET as performed in current clinical practice.

There will be a measurement of CgA levels at baseline (preoperative measures after consent) and afterwards, in 3, 6, 12, and 24 months after resection. Immunoradiometric assay (IRMA, normal values: < 100 ng/mL) will be used.

The collection of blood samples will proceed as detailed below:

Extraction of samples for serum collection:

7 ml of blood without anticoagulants will be allowed to sit for 30 min at room temperature before the serum is separated by centrifugation (3500 rpm). The serum will be stored at -20ºC

Assessments: Baseline (preoperative measures after consent), 3,6, 12, and 24 months

Clinical parameters: weight, height, performance status, vital signs including blood pressure, clinical signs and symptoms, survival data

Blood biochemical parameters: Sodium, potassium, calcium, glucose, urea, creatinina, bilirubin, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT).

Computed tomography (CT) : preoperative condition, and 3,6,12,24 months after resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients having differential diagnosis with PNET in preoperative radiologic diagnosis
* Life expectancy is equal or more than 6 months
* whom written informed consent to participate in the study

Exclusion Criteria:

* renal insufficiency
* taking proton pump inhibitor
* cardiac insufficiency grade 3 and 4
* chronic atrophic gastritis.
* multiple endocrine neoplasia or Cushing's syndrome or mixed tumours or pheochromocytoma or medullary thyroid carcinoma.
* previous history of malignant tumour, with the exception of carcinoma in situ of the uterine cervix or non-melanoma skin cancer
* whom cannot be followed up during the study because of psychology or geographic reasons.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of th CgA in the patient with PNET, change from preoperative levels of CgA at 3 months | preoperation, 3 months
  In the PNET group, the plasma level of CgA was regularly measured.

SECONDARY OUTCOMES:
Diagnostic accuracy of th CgA in the patient with disease progression, change from preoperative levels of CgA at 3, 6,12, and 24 months | preoperation, 3 months, 6 months, 12months, 24 months
  In the PNET group, the plasma level of CgA was regularly checked to follow up the status of disease progression.
Disease progression of PNET using CT imaging, change from preoperative imaging of CT at 3, 6,12, and 24 months | preoperation, 3 months, 6 months, 12months, 24 months
  In the PNET group, the CT was regularly checked to follow up the status of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Songcheol Kim, MD PhD, Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: Undecided